CLINICAL TRIAL: NCT04005664
Title: Prophylactic Phenylephrine and Fluid Co-administration to Reduce Spinal Hypotension During Elective Caesarean Section in a Resource-limited Setting: a Prospective Alternating Intervention Study
Brief Title: Prophylactic Phenylephrine Co-administration During Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE616/17
Record Dates: First submitted 2019-06-19; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Cesarean Section Complications; Anesthesia Complication
MeSH Terms: interventions — Phenylephrine

STUDY DESIGN:
Intervention Model Description: Single centre prospective alternating intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus group (No Intervention): Hypotension occurring under spinal anaesthesia (SBP < 90mmHg) requires pharmacological treatment. The pharmacological management of hypotension, once diagnosed, will be the same regardless of the protocol being used. If the heart rate is greater than 70 beats per minute, phenylephrine will be administered in a dose of 50-100 mcg as an intravenous bolus. If the heart rate is less than 70 beats per minute, ephedrine will be administered in a dose of 5-10 mg. The dose within this range will be decided by the attending anaesthetist. In both arms, Ringers Lactate fluid should run fast if hypotension occurs.
- Phenylephrine coload group (Active Comparator): Phenylephrine 500ug will be added to the first litre of ringer's lactate infused on initiation of spinal anaesthesia. If the phenylephrine infusion protocol is being used, and the mean arterial pressure (MAP) rises to greater than 20% of the initial MAP, and where this rise in MAP is not due to a recent bolus of either phenylephrine or ephedrine (within 2 minutes), the Ringers Lactate infusion will be switched off. The pharmacological management of hypotension, once diagnosed, will be the same regardless of the protocol being used. If the heart rate is greater than 70 beats per minute, phenylephrine will be administered in a dose of 50-100 mcg as an intravenous bolus. If the heart rate is less than 70 beats per minute, ephedrine will be administered in a dose of 5-10 mg. In both arms, Ringers Lactate fluid should run fast if hypotension occurs.
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine — Prophylactic phenylephrine infusion as part of fluid coload
  Other Names: Phenylephrine coload
  Arms: Phenylephrine coload group

SUMMARY:
This single centre prospective alternating intervention study will aim to compare prophylactic phenylephrine given in the first litre of Ringers lactate as co-load in healthy patients having an elective caesarean section under spinal anaesthesia at Edendale Hospital to the existing national protocol guideline - for the treatment of obstetric spinal hypotension.

DETAILED DESCRIPTION:
Spinal anaesthesia is currently standard of care for patients undergoing caesarean section. Obstetric spinal hypotension is a common and important problem, related to important maternal and foetal outcomes. The prevention and treatment of spinal hypotension has been well researched in resource-rich settings, a context different from that encountered in the South African setting. It has been previously shown that a prophylactic phenylephrine infusion is effective in resource-limited settings, but this method is still dependent on the availability of an infusion pump.The ideal dose offering the best risk to benefit profile is 25 to 50 mcg/min. It has recently been shown that a prophylactic phenylephrine infusion, administered by an infusion pump, appears safe and effective in resource-constrained environments. However, some institutions in South Africa are limited by a lack of available infusion pumps. There is an urgent need to translate these research findings into a pragmatic management strategy that is safe and effective where this equipment is lacking. A 18g Jelco allows flow of approximately 100 ml/min in the absence of a pressure bag: therefore with 500 mcg in 1000 ml of ringers lactate and a fully opened line, a maximum dose of 50 mcg.min-1 will be achieved. If the rate is 50 ml/min (20 minutes for the first litre) the dose will be 25 mcg.min-1. This dose range will offer maximum benefit with low risk of side effects.

This exploratory study will establish if a phenylephrine (500 mcg) bolus, added to the first litre of Ringers lactate given as a co-load, is an effective and safe means to prevent post obstetric spinal hypotension. This regime will be compared to the existing South African national protocol of the management of obstetric spinal hypotension. The findings of this study will provide valuable information regarding a safe and potentially effective means to prevent obstetric spinal hypotension.

ELIGIBILITY:
Inclusion Criteria:

* All ASA 1-2 patients undergoing elective caesarean

Exclusion Criteria:

* ASA grade >2 Hypertensive disease in pregnancy Dysrhythmia Failed spinal requiring conversion to a general anaesthetic

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Post spinal hypotension | from insertion of spinal anaesthesia until the delivery of the baby
  The incidence of post spinal hypotension (SBP <90 mmHg)

SECONDARY OUTCOMES:
Maternal symptoms | time of spinal insertion till delivery of the baby
  nausea, vomiting, headache and dizziness.
Maternal cardiac arrest | time of spinal insertion till delivery of the baby
  Requirement for cardiopulmonary resuscitation
Maternal bradycardia | time of spinal insertion till delivery of the baby
  maternal bradycardia requiring atropine administration
Requirement for vasopressor | time of spinal insertion till delivery of the baby
  Number of vasopressor boluses
Highest blood pressure | time of spinal insertion till delivery of the baby
  Highest systolic blood pressure (mmHg)
Lowest blood pressure | time of spinal insertion till delivery of the baby
  Lowest systolic blood pressure (mmHg)
Lowest maternal heart rate | time of spinal insertion till delivery of the baby
  Lowest heart rate (beats per minute)

CONTACTS AND LOCATIONS:
Overall Officials: David G Bishop, PhD, Principal Investigator — University of KwaZulu
Locations (1):
- Edendale Hospital, Pietermaritzburg, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No
No sharing plans

REFERENCES:
- [Result] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Result] Bishop DG, Rodseth RN, Dyer RA. Recipes for obstetric spinal hypotension: The clinical context counts. S Afr Med J. 2016 Aug 1;106(9):861-4. doi: 10.7196/SAMJ.2016.v106i9.10877. PMID 27601104
- [Result] Bishop DG, Cairns C, Grobbelaar M, Rodseth RN. Prophylactic Phenylephrine Infusions to Reduce Severe Spinal Anesthesia Hypotension During Cesarean Delivery in a Resource-Constrained Environment. Anesth Analg. 2017 Sep;125(3):904-906. doi: 10.1213/ANE.0000000000001905. PMID 28244952
- [Result] Allen TK, George RB, White WD, Muir HA, Habib AS. A double-blind, placebo-controlled trial of four fixed rate infusion regimens of phenylephrine for hemodynamic support during spinal anesthesia for cesarean delivery. Anesth Analg. 2010 Nov;111(5):1221-9. doi: 10.1213/ANE.0b013e3181e1db21. Epub 2010 May 21. PMID 20495139